

# Online Survey Informed Consent Form Study Title: A Survey of the Behavior and Experiences of Indoor Tanners

You are being asked to participate in a research study that is being conducted by Dr. Jerod Stapleton, Ph.D. at Rutgers University.

#### **Purpose of the study:**

The purpose of this voluntary research study is to conduct an online survey study to explore beliefs and behaviors related to indoor artificial ultraviolet tanning. Indoor tanning is defined as using tanning beds that use ultraviolet light bulbs to produce tans. You will be one of approximately 500 participants.

#### What will be done?

You will complete a survey, which will take approximately 15 to complete. The survey includes questions about your indoor tanning behavior and how you feel about indoor tanning. Participation in this survey study is voluntary. The only alternative to this study is not to participate.

## **Risks or discomforts:**

Minimal risks are anticipated from taking part in this study. There is always the possibility of tampering from an outside source when using the Internet for collecting information. The confidentiality of your responses will be protected once the data are downloaded from the Internet but there is always a possibility of hacking or other security breaches that could threaten survey confidentiality. Please know that you are free to decide not to answer any question. If you feel uncomfortable or upset with a question, you can skip that question or withdraw from the study altogether.

#### **Benefits of this study:**

There is no direct benefit to you for participating in this study. You will be contributing to knowledge about the health behaviors and experiences of young adults.

#### **Confidentiality:**

Your responses to the online survey will be kept strictly confidential. All efforts will be made to keep your personal information in your research record confidential. Data delivered to the researchers will not contain any personally identifiable information. Your identity will not be released in any publications or reports about this research. No one outside of the research team will know your identity and we will not release your identity in any publications or reports about this research. We have taken the following steps to protect your identity as a research participant:

- The use of Ipsos Public Affairs (formerly GfK Custom Research) online survey software that utilizes secure encryption of data.
- All data from the surveys will be stored in password-protected file and your name and any other identifiable information will not be provided to the investigators from Ipsos Public Affairs.

#### **Compensation:**

You will be provided with the standard compensation for surveys of this type.

#### Withdrawal:

Your participation is voluntary; you are free to withdraw your participation from this study at any time. If you do not want to continue, you can simply leave this website. You also may choose to skip any questions that you do not wish to answer.

## **How the findings will be used:**

Your data may be used in scientific publications and presentations. If the findings from the study are published, you will not be identified by name. Your identity will be kept confidential.

1 Version #: 3 10.25.18





## **Contact information:**

If you have concerns or questions about this research study, please contact the PI (Jerod Stapleton) at (732)-235-8112.

If you have questions about your rights as a research subject, please contact the New Brunswick/Piscataway IRB Director at (732)-235-9806.

#### AGREEMENT TO PARTICIPATE

By beginning the survey, I acknowledge that I am 18 years of age or older, have read this consent form, and agree to take part in the research, with the knowledge that I am free to withdraw my participation at any time without penalty.

